CLINICAL TRIAL: NCT02174133
Title: Impact of LVAD Implantation on Micro- and Macrovascular Function
Acronym: LVAD
Status: Completed | Type: Observational
Sponsor: Klinik für Kardiologie, Pneumologie und Angiologie (Other)
Responsible Party: Sponsor-Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Division of Cardiology, Pulmonary Diseases, Vascular Medicine, Heinrich-Heine University, Duesseldorf
Organization: Heinrich-Heine University, Duesseldorf (Other)
Other Study IDs: LVAD
Record Dates: First submitted 2014-06-24; First posted 2014-06-25 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: End Stage Heart Failure
Keywords: left ventricular assist device; endothelial function; microvascular perfusion; microparticles

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- patients after HTX
- patients after LVAD implantation
- patients with coronary heart disease
- healthy volunteers

SUMMARY:
End stage heart failure is characterized by a critical inability of the heart to meet the organism's blood demand even under resting conditions. Heart transplantation (HTx) is the established therapeutic approach in the treatment of end stage heart failure and still the gold standard treatment. Left ventricular assist devices (LVADs) are considered as a vital therapeutic option to temporarily or permanently assist the failing circulation. The hemodynamic vascular consequences of implanting LVADs have not been studied in detail. The aim of the study is to investigate the effect of LVAD implantation compared to heart transplant (HTx) on micro- and macrovascular function in patients with end stage heart failure.

ELIGIBILITY:
Inclusion Criteria:

* patients after HTX
* patients after LVAD implantation
* patients with stable coronary heart disease and normal systolic left ventricular function
* healthy volunteers
* written informed consent

Exclusion Criteria:

* acute inflammation
* cardiac arrhythmia
* renal failure
* malignant disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with end stage heart failure
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Macrovascular function measured by flow-mediated vasodilation (FMD) | 3 months after implantation

SECONDARY OUTCOMES:
Microvascular function assessed by non-invasive laser Doppler imaging | 3 months after implantation
microparticles determined by Flow Cytometry | 3 months after implantation

CONTACTS AND LOCATIONS:
Overall Officials: Christian Heiss, MD, Principal Investigator — Division of Cardiology, Pulmonology and Vascular Medicine
Locations (1):
- Division of Cardiology, Pulmonology and Vascular Medicine Duesseldorf,, Düsseldorf, Germany